CLINICAL TRIAL: NCT02408510
Title: Pilot Project to Examine the Effects of Exercise on Nocturnal Lipolysis in Men and Women
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 13-0359
Record Dates: First submitted 2015-03-30; First posted 2015-04-03 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: Volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this proof of concept/feasibility study is to use rigorous methodology to explore links between daytime energy status and nocturnal fat metabolism in healthy adults.

DETAILED DESCRIPTION:
This primary goal of this pilot project is to obtain preliminary data demonstrating the feasibility of measuring lipolysis and fat oxidation during sleep in adult human subjects using microdialysis, stable isotope labeling techniques, and whole-room indirect calorimetry. The results of this study will be used in grant applications to perform definitive studies using these methods. The long term goal of this line of research is to explore the mechanisms responsible for sex based differences in the effectiveness of physical activity as an approach to weight loss. Previous longitudinal data have shown that in normal weight and obese individuals, for any given increase in physical activity, there is a significantly greater loss of fat mass in men relative to women [Westerterp, 1997]. These data need to be reconciled, however, with the wealth of data demonstrating that during exercise, women release and oxidize fat more readily than men [Horton, 2009; Horton 1998, Moro 2007]. This phenomenon seems counterintuitive, given that men have less body fat than women and are able to lose more body fat than women when beginning a weight loss program [Bjorntorp, 2007]. Recent data suggests a mechanism to explain this paradox. Specifically, in obese subjects, 24-hour fat oxidation increased following a daytime bout of exercise, and this increase occurred in men only and was driven by a significant increase in fat oxidation not during the day but rather during sleep the night following exercise [Bergouignan, 2014]. Since the predominant source of fuel during sleep is free fatty acids (FFA) released from adipose tissue (i.e., lipolysis), it may be that enhanced sleeping lipolysis is a key factor in how exercise stimulates fat oxidation and thus greater fat loss in males vs. females over time.

The primary objective of the proposed study is to demonstrate the feasibility of measuring nocturnal whole-body and regional lipolysis by using stable isotope techniques and microdialysis of subcutaneous abdominal adipose tissue respectively with the long term goal of determining the effects of acute exercise during the daytime on rates of lipolysis at night in men and women. A secondary objective of this study is to determine if nocturnal regional lipolysis measured by microdialysis of subcutaneous abdominal adipose tissue and whole body lipolysis measured by a stable glycerol isotope infusion are related to dietary and whole body fat oxidation measured by stable isotope labelled fatty acid and whole-room calorimetry, respectively. Finally, the study aims to determine if sleep quality parameters measured by EEG and wrist actigraphy correlate with measures of nocturnal fat oxidation and lipolysis (regional and whole body)

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, 20-35 years of age
* Sedentary (planned exercise < 3 d/week, < 30 min/session)
* Lifetime maximum BMI of 30 kg/m2
* Weight stable by self-report for at least 2 mo before the study (<5% weight change)
* Habitual sleeping pattern of >7 hours not to exceed 9.25 hours of sleep per night
* Zero to low-moderate caffeine intake (not to exceed 500 mg/d)
* Alcohol use fewer than two standard drinks per day per week for males and one or less drinks per day per week for females.

Exclusion Criteria:

* Current smoker
* Use of any medication that could affect lipid metabolism, insulin signaling, or sleep
* Pregnant women will not be enrolled in the study
* Current or chronic medical/psychiatric conditions
* Shift work or dwelling below Denver altitude (1,600 m) a year prior to testing
* Travel across more than one time zone 3 wk before study
* Abnormal eating patterns identified by interview and eating questionnaire
* Screening positive for illicit drugs
* Chronic health conditions such as diabetes,
* Hyper or hypothyroidism
* Sleep apnea (Apnea-Hypopnea Index >5)
* Renal or liver disease, anemia, or cancer
* Regularly go to sleep after midnight
* One or more of the following out-of-range values measured on a fasting blood sample:

  * glucose > 110 mg/dl,
  * thyroid stimulating hormone <0.5 or >5.0 uU/ml,
  * hemoglobin < 14.5 g/dl men, <12.3 g/dl women,
  * alanine amino transferase > 47 U/l,
  * aspartate aminotransferase > 47 U/l,
  * alkaline phosphatase <39 or >117 U/l, or
  * creatinine >1.1 mg/dl.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Adults
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Lipolysis | Overnight (2200h-0700h)
  Measured using stable isotope tracers and microdialysis
Change in Substrate Oxidation | 24 hours
  Measured using whole-room calorimetry

SECONDARY OUTCOMES:
Change in Sleep Quality | Overnight (2200h-0700h)
  Measured using wrist actigraphy
Change in Lipolytic Hormones | Overnight (2200h-0700h)
  Frequent blood sampling to measure growth hormone, cortisol, catecholamines, and other lipolytic hormones

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bessesen, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Westerterp KR, Goran MI. Relationship between physical activity related energy expenditure and body composition: a gender difference. Int J Obes Relat Metab Disord. 1997 Mar;21(3):184-8. doi: 10.1038/sj.ijo.0800385. PMID 9080256
- [Background] Horton TJ, Dow S, Armstrong M, Donahoo WT. Greater systemic lipolysis in women compared with men during moderate-dose infusion of epinephrine and/or norepinephrine. J Appl Physiol (1985). 2009 Jul;107(1):200-10. doi: 10.1152/japplphysiol.90812.2008. Epub 2009 Apr 30. PMID 19407251
- [Background] Horton TJ, Pagliassotti MJ, Hobbs K, Hill JO. Fuel metabolism in men and women during and after long-duration exercise. J Appl Physiol (1985). 1998 Nov;85(5):1823-32. doi: 10.1152/jappl.1998.85.5.1823. PMID 9804587
- [Background] Moro C, Pillard F, de Glisezinski I, Crampes F, Thalamas C, Harant I, Marques MA, Lafontan M, Berlan M. Sex differences in lipolysis-regulating mechanisms in overweight subjects: effect of exercise intensity. Obesity (Silver Spring). 2007 Sep;15(9):2245-55. doi: 10.1038/oby.2007.267. PMID 17890493
- [Background] Bjorntorp PA. Sex differences in the regulation of energy balance with exercise. Am J Clin Nutr. 1989 May;49(5 Suppl):958-61. doi: 10.1093/ajcn/49.5.958. No abstract available. PMID 2655420
- [Background] Bergouignan A, Kealey EH, Schmidt SL, Jackman MR, Bessesen DH. Twenty-four hour total and dietary fat oxidation in lean, obese and reduced-obese adults with and without a bout of exercise. PLoS One. 2014 Apr 8;9(4):e94181. doi: 10.1371/journal.pone.0094181. eCollection 2014. PMID 24714529